CLINICAL TRIAL: NCT04670822
Title: Postpartum Smoking Relapse Prevention by Breastfeeding Promotion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Xiaozhong Wen, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MODCR00004712; R21HD091515 (NIH)
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Results first posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Smoking, Cigarette; Breastfeeding
Keywords: Postpartum; Relapse
MeSH Terms: conditions — Cigarette Smoking; Breast Feeding; Recurrence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breastfeeding intervention group (Experimental): A multicomponent behavioral intervention to promote breastfeeding
  Interventions: Behavioral: Breastfeeding promotion
- Attention placebo control group (Placebo Comparator): General infant care counseling and support
  Interventions: Behavioral: Attention placebo control

INTERVENTIONS:
Behavioral: Breastfeeding promotion — The intervention group will receive multicomponent interventions consisting of 7 half-hour postnatal visits for lactation counseling, family/peer/employer support, contingent financial incentives, and early limited formula milk via syringe (optional for at-risk infants).
  Arms: Breastfeeding intervention group
Behavioral: Attention placebo control — The attention placebo control group will complete the same frequency and duration of study visits as the intervention group but focus on general infant care counseling and support.
  Arms: Attention placebo control group

SUMMARY:
This is a randomized controlled trial to prevent postpartum smoking relapse by breastfeeding promotion. The intervention group (N=30) will receive multicomponent breastfeeding intervention from late pregnancy to 6 months postpartum, while the attention placebo control group (N=30) will receive general infant care counseling and support. The key outcome is the rate of postpartum smoking relapse.

DETAILED DESCRIPTION:
The investigators propose the first randomized controlled trial to reduce postpartum smoking relapse by breastfeeding promotion from late pregnancy to 6 months postpartum. The investigators will enroll 60 pregnant women who successfully quit smoking within 3 months before or during this pregnancy (<28 weeks). All participants will receive breastfeeding education during late pregnancy. Right after delivery, participants who are still smoking abstinent will be randomized into either the breastfeeding intervention group (N=30) or the attention placebo control group (N=30). The intervention group will receive multicomponent interventions consisting of postnatal lactation counseling, family/peer/employer support, contingent financial incentives, and early limited formula milk via syringe (optional for at-risk infants). The control group will receive counseling and support focusing on general infant care with attention and compensation similar to the intervention group. The primary outcomes are rates of postpartum smoking relapse verified by urine cotinine test.

Specific Aim 1 is to examine the efficacy of breastfeeding promotion intervention on postpartum smoking relapse. Specific Aim 2 is to collect preliminary data regarding potential mediating mechanisms: increases in lactation hormones (plasma oxytocin and prolactin), reductions in stress and negative affect, and enhancing mother-infant bonding and maternal motivation to protect the infant from secondhand smoke exposure. This innovative and feasible pilot study can yield promising preliminary data to strongly support our future application of a NIH R01 grant proposal that has the potential to reduce smoking-related harms to both the mother and the infant, and maximize the protective effects of breastfeeding on infant health and development.

ELIGIBILITY:
Inclusion Criteria:

* Be pregnant or in the first 1 month postpartum
* Be 18 years or older
* Have quit smoking cigarettes during or before this pregnancy
* Be willing to receive infant care and breastfeeding education
* Be able to read, listen, and talk in English

Exclusion Criteria:

* Medical conditions contraindicating breastfeeding such as HIV infection, active tuberculosis, and breast removal
* Current heavy drinking (more than 2 drinks a day)
* Current use of illicit substances
* Being strongly against breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaozhong Wen, Principal Investigator — State University of New York at Buffalo
Locations (1):
- Division of Behavioral Medicine Department of Pediatrics Jacobs School of Medicine and Biomedical Sciences State University of New York at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Breastfeeding Intervention Group | Attention Placebo Control Group
Started | 30 | 30
Completed | 25 | 24
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Breastfeeding Intervention Group | Attention Placebo Control Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 9 | 17
  White | 21 | 20 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Pregnancy status [Count of Participants; unit: Participants] — Pregnancy status is verified through testing the levels of human chorionic gonadotropin (hCG) in urine samples. If the urine hCG level is 20 mIU/mL or higher, the test shows a positive result, indicating pregnancy.
  Participants
    Pregnant | 30 | 30 | 60
    Not pregnant | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting to Breastfeed
Description: During postpartum, mothers report their breastfeeding status (exclusive, mixed with formula, non-breastfeeding) every month until 9 months postpartum. Any breastfeeding is defined as exclusive breastfeeding or mixed-feeding breast milk and formula.
Time Frame: 9 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Breastfeeding Intervention Group | Attention Placebo Control Group
Number analyzed (Participants) | 25 | 24
Participants | 13 | 5

ADVERSE EVENTS:
Time Frame: From enrollment until 9 months postpartum
Arm/Group | Breastfeeding Intervention Group | Attention Placebo Control Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT04670822/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/22/NCT04670822/ICF_001.pdf